CLINICAL TRIAL: NCT01527396
Title: Multi-center Prospective Observational Study for the Validation of Preoperative Low-risk Criteria for Lymph Node Metastasis in Endometrial Cancer
Brief Title: Prospective, Observational Study of Low-risk Criteria for Node Metastasis in Endometrial Cancer
Acronym: PALME
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Korean Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, Sokbom Kang, Director, Gynecologic Oncology Research Div., National Cancer Center, Korea
Other Study IDs: KGOG2015
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; lymph node metastasis; lymphadenectomy; risk criteria
MeSH Terms: conditions — Endometrial Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the efficacy of low risk criteria for lymph node metastasis, that was determined by KGOG-2014 retrospective study, in women with endometrial cancer.

DETAILED DESCRIPTION:
The Korean Gynecologic Oncology Group (KGOG) undertook a multi-center retrospective study to develop a preoperative prediction model for lymph node metastasis in endometrial cancer (KGOG-2014). This retrospective multi-center study showed that the accurate identification of a low-risk group for lymph node metastasis among the patients with endometrial cancer can be achieved with the new criteria using preoperative MRI and serum CA-125 assay. In this study, serum CA125 levels and three MRI parameters (deep myometrial invasion, lymph node enlargement, and extension beyond uterine corpus) were found to be independent risk factors for nodal metastasis. Based on the success of KGOG-2014, Korean Gynecologic Oncology Group initiated this prospective, multi-center observational study to validate our prior prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of endometrial cancer before surgical staging.
* Patients with a preoperative magnetic resonance imaging (MRI) and serum CA-125 within 4 weeks from surgical staging.
* Patients who underwent adequate systemic lymph node dissection during surgical staging.

Exclusion Criteria:

* Patients with a histologic feature suggesting sarcoma or squamous cell carcinoma

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Endometrial cancer patients who undergo surgery including systemic lymph node dissection
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity/Specificity | 2014-12-31
Negative predictive value | 2014-12-31
Diagnostic odds ratio | 2014-12-31

CONTACTS AND LOCATIONS:
Overall Officials: Sokbom Kang, Study Chair — National Cancer Center, Korea
Locations (1):
- Korean Gynecologic Oncology Group, Seoul, Kangnam-gu, South Korea